CLINICAL TRIAL: NCT00999102
Title: Nebivolol Vs. Metoprolol: Comparative Effects on Fatigue and Quality of Life
Brief Title: Nebivolol Versus Metoprolol: Comparative Effects on Fatigue and Quality of Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0901010162
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Hypertension
Keywords: hypertension; beta blockers; Metoprolol; blood pressure, high; antihypertensive agents; vascular resistance; adrenergic beta-receptor blockaders; beta-Adrenergic blockers; beta-Adrenergic Blocking Agents; beta-Adrenergic Receptor Blockaders; beta-Blockers, Adrenergic; Bystolic; Nebivolol; Nebivololum; Nebivololum [Latin]; R65,824; Beloc- Zok; H 93/26 succinate; Metoprolol succinate; Seloken ZOC; Selozok; Spesicor Dos; Toprol XL; Toprol-XL; UNII-TH25PD4CCB
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nebivolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol, followed by Metoprolol (Experimental): Participants first received Nebivolol at a dose of 5 mg daily for 4 weeks, followed by 10 mg daily for another 4 weeks (i.e., weeks 1-8 in total). The participants then received Metoprolol at a dose of 50 mg daily for 4 weeks, followed by 100 mg daily for another 4 weeks (i.e., weeks 9-16 in total).
  Interventions: Drug: Metoprolol; Drug: Nebivolol
- Metoprolol, followed by Nebivolol (Experimental): Participants first received Metoprolol at a dose of 50 mg daily for 4 weeks, followed by 100 mg daily for another 4 weeks (i.e., weeks 1-8 in total). The participants then received Nebivolol at a dose of 5 mg daily for 4 weeks, followed by 10 mg daily for another 4 weeks (i.e., weeks 9-16 in total)
  Interventions: Drug: Metoprolol; Drug: Nebivolol

INTERVENTIONS:
Drug: Metoprolol — Metoprolol 50 mg, Metoprolol 100 mg,
  Other Names: Lopressor, Toprol-XL
Drug: Nebivolol — Nebivolol 5 mg, Nebivolol 10 mg.
  Other Names: Bystolic

SUMMARY:
Beta-blockers are prescribed to millions of people for treatment of hypertension. Fatigue is a recognized and common side effect of beta-blockers that can have significant effects on quality of life. Worse, many people taking a beta-blocker for years are not even aware of the reduction of energy with which they are living.

A new vasodilating beta-blocker, nebivolol, which is approved by the FDA for treatment of hypertension, appears to be far less associated with fatigue than are most currently available beta-blockers. The purpose of this study is to compare nebivolol with the current best-selling beta-blocker, metoprolol, and determine whether there is a significant difference in side effects including fatigue, reduced exertion tolerance, and reduced quality of life.

In this study, 30 subjects will take each of the 2 study drugs for 8 weeks, consisting of 4 weeks at a lower dose, and 4 weeks at a higher dose. All dosages are FDA-approved for treatment of hypertension. Subjects and investigators will not know which drug is being administered until completion of the study. Subjects will undergo a treadmill stress test and will complete fatigue and quality of life questionnaires after each 4 weeks of treatment. An echocardiogram and non-invasive measurement of aortic blood pressure will be performed after 8 weeks on each drug. Also, blood will be drawn and stored for possible measurement of drug levels, after 4 and 8 weeks on each drug. Results on each drug will then be compared. If nebivolol is found to cause significantly less fatigue, it would be of substantial importance to the many millions of people who are on life-long beta-blocker therapy, and are living with reduced energy.

DETAILED DESCRIPTION:
* Hypothesis: the beta-blocker nebivolol is associated with less fatigue than metoprolol, the most widely-prescribed beta-blocker
* Methods: a double-blinded crossover trial comparing nebivolol with metoprolol. Experimental procedures: Subjects will undergo electrocardiogram and routine blood testing, unless such tests have been performed within 6 months and are available for review. Subjects entered into the study will receive each of the two study drugs for 8 weeks. Metoprolol succinate will be given at a dose of 50 mg daily for 4 weeks, then 100 mg daily for 4 weeks. For nebivolol, dosage will be 5 mg daily for 4 weeks and 10mg daily for 4 weeks. Identical-appearing pills will be given, and the drugs will be given in randomized order without a placebo run-in period.

At the end of each 4-week treatment period on each drug, subjects will undergo a treadmill stress test (using the standard Cornell protocol), complete Quality of Life and fatigue questionnaires, and have blood drawn and frozen for later analysis for drug levels.

At the end of 8 weeks of treatment on each drug, subjects will undergo echocardiography and applanation tonometry (non-invasive measurement of aortic blood pressure) to assess heart function.

At the end of the study, the blinded subjects will be asked which of the two study drugs they preferred, and the extent to which their energy differed between the two drugs.

-Rationale: Millions of hypertensive patients are on life-long beta-blocker therapy. In many, it reduces cardiac output and increases peripheral resistance to blood flow (1). It is well-established that beta-blockers cause fatigue in many patients and reduce exertion tolerance. Every physician knows this, and tacitly accepts that many patients are living with this unwelcome side effect.

A new beta-blocker, nebivolol, has the standard beta-blocking effects, but also produces blood vessel relaxation (vasodilation), probably through increased secretion of the vasodilator nitric oxide. Studies indicate that nebivolol, unlike most beta-blockers, does not cause constriction of peripheral blood vessels, and is associated with improved heart function (2). Studies suggest that it is also less likely to cause fatigue (3).

Personal experience is consistent with this, as I have observed marked improvement in energy in patients in whom I have prescribed nebivolol in place of a different beta-blocker. The possibility of placebo effect of course cannot be excluded. Nevertheless, the known hemodynamic differences between nebivolol and other beta-blockers, and the positive clinical experience, warrant formal study to determine whether nebivolol is kinder than other beta-blockers in terms of the important side effect of fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are taking, or are about to begin taking, a beta-blocker, and who have the approved indication of hypertension

Exclusion Criteria:

* Orthopedic ailments that would interfere with performance of treadmill testing
* Stroke or heart attack within the previous 1 year
* Symptomatic coronary disease within the past year (angina, shortness of breath)
* Clinically significant pulmonary disease (e.g. emphysema or asthma).
* Poorly controlled hypertension (blood pressure above 160 systolic or 100 diastolic)
* Patients with contra-indications to taking a beta-blocker (asthma or bradyarrhythmia)
* History of tachyarrhythmia (abnormal rapid heart rate)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel J Mann, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the patient population of the Hypertension Center, and from an announcement at the medical center. Subjects were entered from 10/09 to 9/10, and the final subject completed the protocol in 1/11.
Pre-assignment Details: Subjects who were on anti-hypertensives were instructed to continue their medications. Subjects taking a beta-blocker were instructed to stop them. There was no washout period. Individuals with a contraindication to beta-blockers were excluded. 4 subjects dropped out before starting medication for reasons unrelated to the study.
Period: 4 Weeks at Lower Dose of First Drug
Arm/Group | Nebivolol, Followed by Metoprolol | Metoprolol, Followed by Nebivolol
Started | 16 | 17
Completed | 15 | 16
Not Completed | 1 | 1
Period: 4 Weeks at Higher Dose of First Drug
Arm/Group | Nebivolol, Followed by Metoprolol | Metoprolol, Followed by Nebivolol
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: 4 Weeks at Lower Dose of Second Drug
Arm/Group | Nebivolol, Followed by Metoprolol | Metoprolol, Followed by Nebivolol
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: 4 Weeks at Higher Dose of Second Drug
Arm/Group | Nebivolol, Followed by Metoprolol | Metoprolol, Followed by Nebivolol
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Nebivolol followed by Metoprolol or Metoprolol followed by Nebivolol.
Arm/Group | All Study Participants
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Multidimensional Assessment of Fatigue (MAF) Questionnaire: Global Fatigue Score After 4 Weeks of Treatment on Each Drug/Dose Combination.
Description: A 16 item scale that measures 4 dimensions of fatigue: severity, distress, timing, and degree of interference in activities of daily living.
  Range: 1 (no fatigue) to 50 (extreme fatigue).
Time Frame: After 4 weeks of treatment on each drug/dose combination
Population: All participants who received both interventions and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nebivolol 5 mg for 4 Weeks: 31 subjects received Nebivolol 5 mg daily for 4 weeks.
- Metoprolol 50 mg for 4 Weeks: 31 subjects received Metoprolol 50 mg daily for 4 weeks
- Nebivolol 10 mg for 4 Weeks: 31 subjects received Nebivolol 10 mg daily for 4 weeks.
- Metoprolol 100 mg for 4 Weeks: 31 subjects received Metoprolol 100 mg daily for 4 weeks
Arm/Group | Nebivolol 5 mg for 4 Weeks | Metoprolol 50 mg for 4 Weeks | Nebivolol 10 mg for 4 Weeks | Metoprolol 100 mg for 4 Weeks
Number analyzed (Participants) | 31 | 31 | 31 | 31
units on a scale | 18.5 (11.2) | 18.0 (11.2) | 21.0 (11.8) | 20.3 (11.9)
Statistical Analysis 1: Comparison: Nebivolol 5 mg for 4 Weeks vs Metoprolol 50 mg for 4 Weeks; The null hypothesis is that there is no difference in the Global Fatigue Score after 4 weeks of Nebivolol 5 mg (lower dose) vs. 4 weeks of Metoprolol 50 mg (lower dose); Test type: Superiority; p = 0.67, t-test, 2 sided; Paired t-test was performed since each participant received both interventions in a crossover design; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.86 to 2.86] — Direction of Comparison: Mean Global Fatigue Score for Nebivolol 5 mg minus Mean Global Fatigue Score for Metoprolol 50 mg
Statistical Analysis 2: Comparison: Nebivolol 10 mg for 4 Weeks vs Metoprolol 100 mg for 4 Weeks; The null hypothesis is that there is no difference in the Global Fatigue Score after 4 weeks of Nebivolol 10 mg (higher dose) vs. 4 weeks of Metoprolol 100 mg (higher dose); Test type: Superiority; p = 0.72, t-test, 2 sided; Paired t-test was performed since each participant received both interventions in a crossover design; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-3.17 to 4.55] — Direction of Comparison: Mean Global Fatigue Score for Nebivolol 10 mg minus Mean Global Fatigue Score for Metoprolol 100 mg

2. Primary Outcome: Treadmill Exercise Time After 4 Weeks of Treatment on Each Drug/Dose Combination.
Description: Treadmill Exercise Time After 4 Weeks of Treatment on Each Drug/Dose Combination (in minutes). The Treadmill Test was Performed at the 4-week Visit of Each Drug/Dose Combination.
Time Frame: After 4 weeks of treatment on each drug/dose combination
Population: All participants who received both interventions and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Nebivolol 5 mg for 4 Weeks | Metoprolol 50 mg for 4 Weeks | Nebivolol 10 mg for 4 Weeks | Metoprolol 100 mg for 4 Weeks
Number analyzed (Participants) | 31 | 31 | 31 | 31
minutes | 833.9 (266.1) | 840.9 (288.6) | 841.2 (265.4) | 867.1 (249.8)
Statistical Analysis 1: Comparison: Nebivolol 5 mg for 4 Weeks vs Metoprolol 50 mg for 4 Weeks; The null hypothesis is that there is no difference in Treadmill Exercise Time after 4 weeks of Nebivolol 5 mg (lower dose) vs. 4 weeks of Metoprolol 50 mg (lower dose); Test type: Superiority; p = 0.89, t-test, 2 sided; Paired t-test was performed since each participant received both interventions in a crossover design; Mean Difference (Final Values) = -7.03, 95% CI 2-sided [-108.99 to 94.92] — Direction of Comparison: Mean Treadmill Exercise Time for Nebivolol 5 mg minus Mean Treadmill Exercise Time for Metoprolol 50 mg
Statistical Analysis 2: Comparison: Nebivolol 10 mg for 4 Weeks vs Metoprolol 100 mg for 4 Weeks; The null hypothesis is that there is no difference in Treadmill Exercise Time after 4 weeks of Nebivolol 10 mg (higher dose) vs. 4 weeks of Metoprolol 100 mg (higher dose); Test type: Superiority; p = 0.43, t-test, 2 sided; Paired t-test was performed since each participant received both interventions in a crossover design; Mean Difference (Final Values) = -25.90, 95% CI 2-sided [-91.55 to 39.75] — Direction of Comparison: Mean Treadmill Exercise Time for Nebivolol 10 mg minus Mean Treadmill Exercise Time for Metoprolol 100 mg

ADVERSE EVENTS:
Time Frame: After 4 weeks on either study drug.
Description: All-Cause Mortality; Serious; Other.
Arm/Group | Nebivolol 5 mg for 4 Weeks | Metoprolol 50 mg for 4 Weeks | Nebivolol 10 mg for 4 Weeks | Metoprolol 100 mg for 4 Weeks
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 1/33 | 1/33 | 0/31 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol 5 mg for 4 Weeks (N=33) | Metoprolol 50 mg for 4 Weeks (N=33) | Nebivolol 10 mg for 4 Weeks (N=31) | Metoprolol 100 mg for 4 Weeks (N=31)
Fatigue (General disorders) | 1 | 1 | 0 | 0 — 1 subject on each drug dropped out of the study with complaint of fatigue. The symptom ceased with discontinuation of the drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No